CLINICAL TRIAL: NCT04167657
Title: A Phase II Single-arm Study of Sintilimab After Thoracic Radiation in Previously Treated Advanced NSCLC
Brief Title: SinTilimab After Radiation (STAR Study)
Acronym: STAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wang mengzhao, Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-1856
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Carcinoma, Non-Small Cell Lung
Keywords: Advanced non-small cell lung cancer; Immunotherapy; Radiation; PD-1; Sintilimab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm1 (Experimental): Sintilimab monotherapy every 3 weeks, after a radiation targeting a single location no less than dose 30Gy( 6 Gy × 5, or other ), or the planned dose could reach 30 Gy.
  Interventions: Drug: Sintilimab

INTERVENTIONS:
Drug: Sintilimab — Sintilimab 200mg IV, every 3 weeks, until progressive disease (PD), intolerable toxicity, or at a maximum of 24 months.
  Before enrollment, patient should undergo radiation no less than dose 30Gy( 6 Gy × 5, or other ), or the planned dose could reach 30 Gy. Sintilimab shall be started no later than 3 weeks after radiation. Radiotherapy can be performed on the same day as sintilimab.

SUMMARY:
This study is a single-arm multi-center phase II clinical study, which aims to investigate the efficacy and safety of sintilimab after radiotherapy in patients with advanced NSCLC who failed first-line or second-line systemic treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent;
2. Age ≥ 18 years ;
3. Histologically or cytologically confirmed NSCLC, without EGFR sensitive mutation (must) or no known ALK/ROS1 positive;
4. Stage IIIB-IV (AJCC 8th edition) or recurrent/progressive disease after multidisciplinary treatment for local advanced disease or chemotherapy intolerant patients;
5. Patients must have disease progression or recurrence after receiving first/second line systemic therapy for advanced or metastasis disease, or patients with chemotherapy intolerance during chemotherapy: 1) Maintenance therapy after platinum based chemo-doublet shall not be considered as a separated treatment regimen, 2)Patients with locally advanced disease treated with platinum-based adjuvant, neoadjuvant therapy or radical chemoradiotherapy, and tumor recurrence ( local or metastatic ) within 6 months after completion of treatment are suitable for inclusion; 3) Subjects who relapsed more than 6 months after receiving platinum-based adjuvant, neoadjuvant therapy or radical chemoradiotherapy for locally advanced disease, and then progressed during or after receiving systemic treatment for recurrent tumors were suitable for inclusion; 4) Patients who received platinum-based double-drug chemotherapy after progression or chemotherapy intolerance were considered as second-line patients after first-line treatment; 5) After the progression of platinum-containing double-drug chemotherapy, patients who progressed again with a single-drug chemotherapy regimen or chemotherapy intolerance were considered as third-line patients after second-line treatment.
6. ECOG PS 0-1, with expected survival over 3 months;
7. Patients shall have at least one leision eligible for radiation, e.g. bone metastasis, intrapulmonary node, adrenal disease, etc. Patient must have at least one disease (other than radiation target) according to RECIST 1.1: 1) Patient must have received radiation for 1 location after disease progression or recurrence after first line treatment for advanced or metastasis disease, the biological dose of a single site of radiotherapy is required to exceed 30 Gy ( 6 Gy × 5, or other ) or the plan can reach 30 Gy. 2) Radiotherapy can be performed on the same day as Sindilizumab, but the last radiotherapy is no more than 3 weeks after the start of Sindilizumab treatment.
8. Adequate marrow and organ function as per baseline CBC/CMP/Urine test;
9. Prior systemic anti-tumor therapy should be completed at least 4 weeks before enrollment, and adverse events of prior treatment shall be return to ≤G1 per CTCAE (except for alopecic or any non-clinical significant laboratory abnormalities) ;
10. Women with childbearing potential or men whose female partners are with childbearing potential must agree to use efficient contraceptive methods during the study treatment period until 90 days after last dose of study treatment.

Exclusion Criteria:

1. Previously treated by any immune therapy;
2. Active infection including HBV, HCV, and HIV;
3. Serious marrow or organ malfunction, e.g. hepatic or renal dysfunction;
4. Patients with unstable CNS metastasis or require corticosteroids to control CNS symptoms. Patients with stable brain metastasis after radiation (3 weeks) will be eligible;
5. Active or autoimmune disease;
6. ILD, including drug-induced ILD, radiation pneumonia that required corticosteroids, or any clinical implication for active ILD;
7. Any course that lead to treatment with continuous systemic corticosteroids >10 mg/day prednisone or equivalent dose of other steroids;
8. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Time Frame: up to 12 months after enrollment or study close
  ORR (per RECIST 1.1 as assessed by the investigator) is defined as the proportion of patients with a complete response (CR) or partial response (PR) as their best respons ORR (per RECIST 1.1 as assessed by the investigator) is defined as the proportion of patients with a complete response (CR) or partial response (PR) as their best respons

CONTACTS AND LOCATIONS:
Overall Officials: Mengzhao Wang, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Department of Respiratory Medicine, Peking Union Medical College Hospita, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Undecided